CLINICAL TRIAL: NCT03755713
Title: A Phase 1, Randomized, Placebo-Controlled Study to Evaluate Safety, Tolerability and Immune Response in Adolescents Allergic to Peanut After Receiving Intradermal Administration of ASP0892 (ARA-LAMP-vax), a Single Multivalent Peanut (Ara h1, h2, h3) Lysosomal Associated Membrane Protein DNA Plasmid Vaccine
Brief Title: A Study to Evaluate Safety, Tolerability and Immune Response in Adolescents Allergic to Peanut After Receiving Intradermal Administration of ASP0892 (ARA-LAMP-vax), a Single Multivalent Peanut (Ara h1, h2, h3) Lysosomal Associated Membrane Protein DNA Plasmid Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0892-CL-1002
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Peanut Allergy
Keywords: ASP0892; Peanut Allergy
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ASP0892 Low Dose (Cohort A) (Experimental): Each cohort will consist of 10 participants (ASP0892 n = 8 and placebo n = 2). The data will be assessed by the Data Monitoring Committee (DMC) after all enrolled cohort A participants complete visits through day 43. Assessments for safety, tolerability, and dose escalation will occur prior to beginning cohort B.
  Interventions: Drug: ASP0892
- ASP0892 High Dose (Cohort B) (Experimental): After all participants in cohort A complete study procedures, the DMC will review the safety and tolerability data and provide recommendations depending on the nature, frequency and severity of the safety profile reviewed. Recommendations will be to proceed with escalation to the next higher dose or stop dose escalation (i.e., no further dosing with study drug).
  Interventions: Drug: ASP0892
- Placebo (Placebo Comparator): Each cohort will consist of 10 participants (ASP0892 n = 8 and placebo n = 2). The data will be assessed by the Data Monitoring Committee (DMC) after all enrolled cohort A participants complete visits through day 43. Assessments for safety, tolerability, and dose escalation will occur prior to beginning cohort B.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP0892 — Intradermal
  Arms: ASP0892 High Dose (Cohort B); ASP0892 Low Dose (Cohort A)
Drug: Placebo — Intradermal; normal saline solution
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of ASP0892 after intradermal (ID) injection in adolescent participants with peanut allergy.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index (BMI) ≥ 3rd percentile and ≤ 97th percentile.
* Subject has a physician-diagnosed peanut allergy or history of peanut allergy. Subjects with history of nonsevere anaphylaxis (Grade ≤ 3) to peanuts (including mild wheezing or dyspnea without hypoxia) will be enrolled.
* Subject has an anti-Ara h2 Immunoglobulin E (IgE) measured by ImmunoCAP > 0.35 kU/L.
* Subject has a positive Skin prick test (SPT) to peanut with a change in wheal diameter ≥ 3 mm as compared to a negative control.
* Subject has a positive peanut Double-blinded placebo-controlled food challenge (DBPCFC) at Screen 2 visit with an eliciting dose ≤ 300 mg peanut protein (≤ 444 mg cumulative reactive dose [CRD]).
* Female subject must either:

  * Be of non-childbearing potential, clearly premenarchal; documented surgically sterile (e.g., hysterectomy, bilateral salpingectomy, bilateral oophorectomy).
  * Or, if of childbearing potential, agrees not to try to become pregnant during the study; and have a negative urine pregnancy test at screening and at day 1 (predose); and if heterosexually active, agrees to consistently use 1 form of highly effective birth control starting at screening and throughout the study period.
* Female subject must agree not to breastfeed starting at screening and throughout the study period, and for 28 days after the final study drug administration.
* Female subject must not donate ova starting at screening and throughout the study period, and for 28 days after the final study drug administration.
* A heterosexually active male subject with female partner(s) who are of childbearing potential is eligible if:

  * Agrees to use a male condom starting at screening and continue throughout study treatment and for 28 days after the final study drug administration. If the male subject has not had a vasectomy or is not sterile, the subjects female partner(s) is utilizing 1 form of highly effective birth control starting at screening and continue throughout study treatment and for 90 days after the male subject receives his final study drug administration.
* Male subject must not donate sperm starting at screening and throughout the study period, and for 90 days after the final drug administration.
* Subject and subject's parent(s) or legal guardian agree that the subject will not participate in another interventional study while participating in the present study.

Exclusion Criteria:

* Subject has severe anaphylaxis to peanuts (Grades 4 or 5 including dyspnea associated with hypoxia, cyanosis, hypotension or neurological compromise) per the Grading of Food-Induced Anaphylaxis According to Severity of Clinical Symptoms based on historical clinical symptoms.
* Subject develops a Grade 4 or 5 reaction during the DBPCFC, per the Grading of Food- Induced Anaphylaxis According to Severity of Clinical Symptoms based on historical clinical symptoms.
* Subject has received or is planning to receive administration of any vaccine (other than injectable Influenza vaccine) from 28 days prior to the first dose through 2 weeks after the last dose of the study vaccine.
* Subject received any specific immunotherapy for allergy (e.g., epicutaneous immunotherapy [EPIT], sublingual immunotherapy [SLIT], Subcutaneous immunotherapy [SCIT] and oral immunotherapy [OIT]) during the past 12 months, currently or plans to receive during the course of the study.
* Subject has used the following drug(s) prior to the dosing of the study vaccine:

  * Within 2 months prior to study vaccine administration: Systemic (or inhaled) steroid, chemical mediator-isolation inhibitor, T helper cell type 2 (Th2) cytokine inhibitor, thromboxane A2 synthesis inhibitor, thromboxane A2 receptor antagonist, β-blocker, angiotensin-converting enzyme inhibitors and/or angiotensin-receptor blockers
  * Within 3 months prior to study vaccine administration: Biologics and/or immune modulators (including anti-TNFα antibody and anti-IgE monoclonal antibody)
* Subject has history of allergic reactions such as anaphylactic shock, angioedema with airway constriction or hypotension caused by food other than peanut and/or medical products (including vaccine) in the past.
* Subject's laboratory test results at screening or prior to study drug dosing on day 1 are outside the normal limits and are considered clinically significant.
* Subjects with anti-Lysosomal associated membrane protein (LAMP)-1 antibodies above the cut-point for the Tier 1 assay and who are confirmed positive in the Tier 2 assay at Screen 1 visit (baseline).
* Subject had a positive test result for hepatitis B surface (HBs) antigen, hepatitis C virus (HCV) antibody or human immunodeficiency virus (HIV) antigen/antibody.
* Subject had a positive urine drug screen result.
* Subject has immune disorders (including autoimmune disease) and/or diseases requiring immunosuppressive drugs.
* Subject was diagnosed with immunodeficiency in the past.
* Subject has uncontrolled hypertension.
* Subject has a history of cardiovascular disease, arrhythmias, chronic lung disease, active eosinophilic gastrointestinal disease or any other medical or surgical conditions, which, places the subject at increased risk for participation in the study.
* Subject has a complication or medical history of respiratory disease, which requires medical treatment.
* Subject has a complication or medical history of malignant tumor.
* Subject has mental conditions such as schizophrenia, bipolar disorder, dementia or major depressive disorder.
* Subject has severe or poorly controlled atopic dermatitis or generalized eczema.
* Subject is unable to discontinue antihistamines within 7 days or 5 half-lives (whichever duration is longer) prior to SPT and oral food challenge procedures.
* Subject has asthma other than mild intermittent asthma (National Heart, Lung and Blood Institute [NHLBI] Guidelines, July 2007) and has a forced expiratory volume in 1 second value < 80% and/or requiring chronic maintenance treatment (i.e., inhaled corticosteroids).
* Subject has already received injection of Lysosomal associated membrane protein (LAMP)-vax such as ASP0892.
* Subject has received investigational therapy within 35 days or 5 half-lives, whichever is longer, prior to screening.
* Subject's parent(s) or legal guardian is an employee of the Astellas Group or vendors involved in the study.
* Subject has any condition, which, makes the subject unsuitable for study participation.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2021-10-11 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by Treatment Emergent Adverse Events (TEAEs) | Up to Day 576
  Adverse Events (AEs) will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). AEs starting or worsening after the first dose of study drug up through study completion will be considered treatment-emergent.
Safety as assessed by local reactogenicity reactions | Up to Day 50
  Participants will be asked to record local reactogenicity (pain, tenderness; erythema/redness, Induration/Swelling) on a daily basis for 7 consecutive days after the injection, each treatment will be summarized. Grades range from 1 (mild) to 4 (Potentially Life Threatening).
Safety as assessed by systemic reactogenicity reactions | Up to Day 50
  Participants will be asked to record systemic reactogenicity (nausea/vomiting, diarrhea, headache, fatigue, myalgia) on a daily basis for 7 consecutive days after the injection, each treatment will be summarized. Grades range from 1 (mild) to 4 (Potentially Life Threatening).
Number of participants with vital signs abnormalities and/or adverse events | Up to Day 576
  Number of participants with potentially clinically significant vital sign values.
Number of participants with laboratory value abnormalities and/or adverse events | Up to Day 576
  Number of participants with potentially clinically significant laboratory values.
Safety assessed by Anti-LAMP-1 antibody | Up to Day 576
  Anti-LAMP-1 antibody formation for all participants will be summarized for each treatment by visit using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (7):
- United States (7):
  - Arkansas Children's Hospital Research Institute, Little Rock, Arkansas
  - Sean N Parker Center for Allergy & Asthma Research, LPCH El Camino Hospital, Mountain View, California
  - The University of Chicago Medicine, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Asthma, Inc., Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Ferslew BC, Smulders R, Zhu T, Blauwet MB, Kusawake T, Spence A, Aldridge K, DeBerg HA, Khosa S, Wambre E, Chichili GR. Safety and immunopharmacology of ASP0892 in adults or adolescents with peanut allergy: two randomized trials. Allergy. 2024 Feb;79(2):456-470. doi: 10.1111/all.15931. Epub 2023 Nov 27. PMID 38010254
- See also: Link to results on the Astellas Clinical Study Results website. — https://www.clinicaltrials.astellas.com/study/0892-CL-1002/
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=14536&tenant=MT_AST_9011